CLINICAL TRIAL: NCT04707859
Title: Danish Study of Non-Invasive Diagnostic Testing in Coronary Artery Disease 3
Acronym: Dan-NICAD 3
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: Dan-NICAD 3
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Angina Pectoris; Atherosclerosis; Coronary Artery Disease; Myocardial Ischemia
Keywords: Positron Emission Tomography; Coronary Computed Tomography Angiography; Rubidium; 15O water; Fractional flow reserve
MeSH Terms: conditions — Angina Pectoris; Atherosclerosis; Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — From all participants consenting to the study, blood samples are drawn prior to CCTA contrast administration. Samples are centrifuged and processed into etylen-diamin-tetra-eddikesyre (EDTA) and heparin treated plasma, and serum, which are aliquoted into individual matrix tubes and placed at -20°C. In addition, one blood samples are placed directly in the freezer for later extraction of genomic DNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: Participants consenting to the study will undergo:
  a1) An interview a2) Blood samples withdrawals a3) ECG a4) Non-enhanced CT a5) CCTA a6) Follow-up for > 10 years
  Patients with suspicion of coronary stenosis detected by CCTA will after undergo:
  b1) Rb PET b2) 15O-water PET b3) Invasive coronary angiography with 3 vessel measurement of fractional flow reserve (FFR), coronary flow reserve (CFR) and index of microvascular resistance (IMR)
  Interventions: Diagnostic Test: Head to head comparison: Rubidium vs 15O-water PET

INTERVENTIONS:
Diagnostic Test: Head to head comparison: Rubidium vs 15O-water PET — Head to head comparison with invasive FFR as reference. Adjustment for abnormal microcirculation

SUMMARY:
In a cohort of symptomatic patients referred to coronary computed tomography angiography (CCTA), the investigators aim is:

1. To investigate and compare the diagnostic precision of Rubidium Positron Emission Tomography (Rb PET) and 15O-water PET (15O-water PET) in patients where CCTA does not exclude obstructive coronary artery disease (CAD) using invasive coronary angiography with fractional flow reserve (ICA-FFR) as reference standard.
2. To study the diagnostic accuracy and prognostic value of computed tomography fractional flow reserve (CT-FFR) in patients where CCTA does not exclude obstructive CAD with ICA-FFR as reference standard.
3. To validated a pre-test probability model including genetic and circulating biomarkers.
4. To identify and characterize genetic risk variants and circulating biomarkers importance in developing CAD.
5. To evaluate the bone mineral density in the hip and spine and correlate this to the degree of vascular calcification.

DETAILED DESCRIPTION:
CCTA has become the preferred diagnostic modality for symptomatic patients with low to intermediate risk of CAD. Of the patients examined, CCTA exclude cardiovascular disease in 70-80% with an excellent negative predictive value of more than 95%. Having a low positive predictive value, however, CCTA often overestimates the severity of CAD, especially in patients with moderate to severe coronary calcification. Following CCTA, patients are hence unnecessarily tested using golden standard ICA-FFR. These ICAs often show no obstructive coronary stenosis and are therefore not followed by revascularization. The issues outlined raises the question of whether it is possible (1) to make a more precise risk stratification and consequently better selection of patients prior to CCTA and (2) to reduce the number of patients referred for unnecessary ICAs following CCTA.

In patients with suspicion of coronary stenosis detected by CCTA, current guidelines recommend verification of myocardial ischemia. Dan-NICAD 3 investigate the diagnostic accuracy of advanced non-invasive myocardial perfusion imaging tests; Rb PET and 15O-water PET. These examinations have shown a high diagnostic accuracy in symptomatic patients with high risk of ischemic heart disease. However, the diagnostic accuracy is not investigated in patients as follow-up after CCTA. In addition, microcirculation may impact the correlation between PET and ICA-FFR which this study will investigate further.

An alternative way to increase the diagnostic accuracy of CCTA and thus avoid unnecessary downstream testing using ICA is to utilize the ability to extract physiological information from the anatomical CCTA images. CT-FFR has in previous studies shown promising results. In addition, calculated estimation of microcirculatiory function is under development and this study will validated these algorithms. Furthermore, the prognostic value of CT-FFR is unknown and will be tested in the pooled cohort of Dan-NICAD 1, 2 and 3.

Obtained during ICA, quantitative flow ratio (QFR) is a novel wire-free approach for fast computation of FFR with potential to increase the global use of physiological lesion assessment. QFR is superior to traditional assessment of intermediate coronary lesions based on quantitative coronary analysis of ICA. However, disagreement between ICA-FFR and QFR has been identified in up to 20% of all measurements. QFR will be validated compared to PET and ICA-FFR.

ELIGIBILITY:
- Inclusion Criteria:

Patients with an indication for CCTA. Qualified patients who have signed a written informed consent form.

- Exclusion Criteria:

Demography and co-existing cardiac morbidity specific: Age below 30 years, patients having a donor heart, a mechanic heart, or mechanical heart pump, suspicion acute coronary syndrome or previous revascularization.

CCTA: Pregnant women, including women who are potentially pregnant or lactating, reduced kidney function, with an estimated glomerular filtration rate (eGFR) < 40 mL/min or allergy to X-ray contrast medium.

PET: contra-indication for adenosine (severe asthma, advanced atrioventricular block, or critical aorta stenosis).

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an indication for CCTA.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-01-05 (Actual); Primary Completion 2022-07-05 (Estimated); Study Completion 2023-01-05 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of Rb PET and 15-O PET | ICA: 4 weeks after inclusion
  Head-to-head comparison using ICA-FFR as reference standard stratified for CFR

SECONDARY OUTCOMES:
Diagnostic accuracy of QFR vs. ICA-FFR | ICA: 4 weeks after inclusion
  Head-to-head comparison using ICA-FFR as reference standard
Pre-test probability model of CAD | ICA: 4 weeks after inclusion
  Advanced pre-test probability model of CAD included clinical information, genetic and circulating biomarkers
Diagnostic accuracy of QFR | ICA: 4 weeks after inclusion
  Head-to-head comparison using ICA-FFR as reference standard
Diagnostic accuracy of CT-FFR | ICA: 4 weeks after inclusion
  Head-to-head comparison with PET using ICA-FFR as reference standard
Effect of reduced myocardial perfusion defect on symptoms of angina pectoris | Re-PET: 12 months after inclusion
  12 months re-PET investigation will by used for estimation of reduction of myocardial perfusion defect size which will be correlated with symptoms of angina pectoris 3 and 12 mdr. after ICA
Prognostic value of clinical, biomarker, genetic information | Follow-up: Myocardial infarction and mortality rates after 3+5+10 years
  Prognotic models will be developed based on machine learning algorithms
Prognostic value of clinical markers, CCTA, Rb PET, 15O-water PET, CT-FFR and QFR | Follow-up: Myocardial infarction and mortality rates after 3+5+10 years
  Prognotic models will be developed based on machine learning algorithms
Predictive models of obstructive CAD | ICA: 4 weeks after inclusion
  Development of pre-test probability models of obstructive CAD at ICA

CONTACTS AND LOCATIONS:
Overall Officials: Simon Winther, MD, PhD, Principal Investigator — Hospital Unit West, Herning, Denmark
Locations (1):
- Gødstrup Hospital, Herning, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nissen L, Winther S, Isaksen C, Ejlersen JA, Brix L, Urbonaviciene G, Frost L, Madsen LH, Knudsen LL, Schmidt SE, Holm NR, Maeng M, Nyegaard M, Botker HE, Bottcher M. Danish study of Non-Invasive testing in Coronary Artery Disease (Dan-NICAD): study protocol for a randomised controlled trial. Trials. 2016 May 26;17(1):262. doi: 10.1186/s13063-016-1388-z. PMID 27225018
- [Background] Rasmussen LD, Winther S, Westra J, Isaksen C, Ejlersen JA, Brix L, Kirk J, Urbonaviciene G, Sondergaard HM, Hammid O, Schmidt SE, Knudsen LL, Madsen LH, Frost L, Petersen SE, Gormsen LC, Christiansen EH, Eftekhari A, Holm NR, Nyegaard M, Chiribiri A, Botker HE, Bottcher M. Danish study of Non-Invasive testing in Coronary Artery Disease 2 (Dan-NICAD 2): Study design for a controlled study of diagnostic accuracy. Am Heart J. 2019 Sep;215:114-128. doi: 10.1016/j.ahj.2019.03.016. Epub 2019 May 1. PMID 31323454
- [Derived] Westra J, Rasmussen LD, Karim SR, Jensen RV, Ejlersen JA, Gormsen LC, Bottcher M, Eftekhari A, Winther S, Christiansen EH. Coronary microvascular disease in patients referred to coronary angiography following coronary computed tomography angiography. EuroIntervention. 2025 Sep 1;21(17):e1005-e1014. doi: 10.4244/EIJ-D-24-01155. PMID 40887988
- [Derived] Rasmussen LD, Sikjaer M, Soby JH, Pedersen OB, Westra J, Efthekhari A, Christiansen EH, Foldyna B, Williams MC, Dweck MR, Newby DE, Douglas PS, Bottcher M, Winther S. Dual probability approach for risk adjustment in patients with a low clinical likelihood of coronary artery disease. Eur Heart J Cardiovasc Imaging. 2025 Aug 29;26(9):1507-1517. doi: 10.1093/ehjci/jeaf193. PMID 40590244
- [Derived] Winther S, Rasmussen LD, Karim SR, Westra J, Dahl JN, Soby JH, Nissen L, Lomstein FB, Wurtz M, Sundboll JM, Ejlersen JA, Mortensen J, Tolbod LP, Sondergaard HM, Hansson NCL, Nyegaard M, Jensen RV, Madsen MA, Christiansen EH, Gormsen LC, Bottcher M. Myocardial Perfusion Imaging With PET: A Head-to-Head Comparison of 82Rubidium Versus 15O-water Tracers Using Invasive Coronary Measurements as Reference. Circ Cardiovasc Imaging. 2025 Jun;18(6):e017479. doi: 10.1161/CIRCIMAGING.124.017479. Epub 2025 Apr 3. PMID 40177753
- [Derived] Brix GS, Rasmussen LD, Rohde PD, Nissen L, Nyegaard M, O'Donoghue ML, Bottcher M, Winther S. Elevated lipoprotein(a) levels are independently associated with the presence of significant coronary stenosis in de-novo patients with stable chest pain. Am Heart J. 2025 Apr;282:103-113. doi: 10.1016/j.ahj.2025.01.001. Epub 2025 Jan 7. PMID 39788470
- [Derived] Rasmussen LD, Westra J, Karim SR, Dahl JN, Soby JH, Ejlersen JA, Gormsen LC, Eftekhari A, Christiansen EH, Bottcher M, Winther S. Microvascular resistance reserve: impact on health status and myocardial perfusion after revascularization in chronic coronary syndrome. Eur Heart J. 2025 Feb 3;46(5):424-435. doi: 10.1093/eurheartj/ehae604. PMID 39217607
- [Derived] Rasmussen LD, Karim SR, Westra J, Nissen L, Dahl JN, Brix GS, Knuuti J, Schmidt SE, Holm NR, Christiansen EH, Eftekhari A, Bottcher M, Winther S. Clinical Likelihood Prediction of Hemodynamically Obstructive Coronary Artery Disease in Patients With Stable Chest Pain. JACC Cardiovasc Imaging. 2024 Oct;17(10):1199-1210. doi: 10.1016/j.jcmg.2024.04.015. Epub 2024 Jul 3. PMID 38970593
- [Derived] Winther S, Dupont Rasmussen L, Westra J, Abdulzahra SRK, Dahl JN, Gormsen LC, Christiansen EH, Brix GS, Mortensen J, Ejlersen JA, Sondergaard HM, Hansson NCL, Holm NR, Knudsen LL, Eftekhari A, Moller PL, Rohde PD, Nyegaard M, Bottcher M. Danish study of Non-Invasive Testing in Coronary Artery Disease 3 (Dan-NICAD 3): study design of a controlled study on optimal diagnostic strategy. Open Heart. 2023 Jul;10(2):e002328. doi: 10.1136/openhrt-2023-002328. PMID 37487656